CLINICAL TRIAL: NCT00512382
Title: The Nature of Reflux-respiratory Symptoms Association in Difficult to Treat Asthmatic/Wheezing Babies Using Impedance and Wheezy Monitoring
Brief Title: The Nature of Reflux-respiratory Symptoms Association in Difficult to Treat Wheezing\Coughing Babies
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Avigdor Mandelberg, Director, Pediatric Pulmonry Unit, Wolfson Medical Center
Other Study IDs: 688 special
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Asthma; Cough; Wheezing
Keywords: GER Gastrointestinal reflux; Aspiration; ASHTMA; COUGH; WHEEZE; PH-IMPEDANCE; WEEM Wheezy Monitor
MeSH Terms: conditions — Asthma; Cough; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Babies and small children 1-24 months
  Interventions: Device: WEEM - Wheezy Monitoring
- B: Children 2-18 years old
  Interventions: Device: WEEM - Wheezy Monitoring

INTERVENTIONS:
Device: WEEM - Wheezy Monitoring — loudspeaker recording (WEEM) is attached externally to the chest simultaneously with PH-Impedance.

SUMMARY:
GER and respiratory symptoms are both common phenomenon in children. Both can coexist in the same patient by chance alone. Research reveals increased incidence for both to coexist leading to suspect a temporal association and possible causality. Therefore we conducted an observational study To determine the primary cause (RS or GER)using for the first time both PH-Impedance as measurements of GER and Wheezy monitoring (WEEM) that records simultaneously wheeze and cough noises. Both modalities will be recorded for 12-24 hours. If GER precedes cough/wheeze recordings it points to GER being the possible precipitating factor and vice versa.

DETAILED DESCRIPTION:
GER and respiratory symptoms are both common phenomenon in children. Both can coexist in the same patient by chance alone. Research reveals increased incidence for both to coexist leading to suspect a temporal association and possible causality. Therefore we conducted an observational study To determine the primary cause (RS or GER)using for the first time both PH-Impedance as measurements of GER and Wheezy monitoring (WEEM) that records simultaneously wheeze and cough noises. Both modalities will be recorded for 12-24 hours. If GER precedes cough/wheeze recordings it points to GER being the possible precipitating factor.However, If cough/wheeze precedes GER recordings it points to cough/wheeze being the possible precipitating factor. The recordings will be investigated 1 minute before and one minute after each event.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month - 18 years old
* Difficult to treat asthma
* Difficult to treat cough
* Difficult to treat other respiratory symptoms

Exclusion Criteria:

* Children on artificial ventilation
* Children not compliant with PH-Metria and/or WEEM

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We studied 23 consecutive Difficult to treat infants and children suspected of suffering from both RS and GER with chronic respiratory symptoms. However, four dropted due to technical problems wiht the equipment. In 19 patients We fully analyzed the respiratory sounds one minute during and one minute before and one minute after each GER episode, and in all parental markings of cough.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Mandelberg, MD, Study Director — Edith Wolfson Medical Center, and Sackler School of Medicine, Tel Aviv University, Tel aviv
Locations (1):
- Wolfson Medical center and Sackler School of Medicine, Tel Aviv University, Tel, Holon, Israel